CLINICAL TRIAL: NCT05600673
Title: Efficacy of Combined CO2 Fractional Laser With Bimatoprost 0.03% in Treatment of Alopecia Areata
Brief Title: Combined CO2 Fractional Laser With Bimatoprost 0.03% Treatment of Alopecia Areata
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ahmed Hassan Nouh MD (Other)
Responsible Party: Sponsor-Investigator, Ahmed Hassan Nouh MD, Lecturer of Dermatology, Venereology and Andrology department, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlAzharUE
Record Dates: First submitted 2022-10-22; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata; Bimatoprost; CO2 Fractional Laser
MeSH Terms: conditions — Alopecia Areata | interventions — Bimatoprost; Solutions

STUDY DESIGN:
Intervention Model Description: In this design, subjects are randomized to 2 study arms and each study arm will be allocated a different intervention. After randomization each participant will stay in their assigned treatment arm for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimatoprost + CO2 (Experimental): Each patient received three CO2 fractional laser sessions 3 weeks apart with immediate and subsequent daily Bimatoprost 0.03%,1 drop for each 1cm².
  Interventions: Drug: Bimatoprost 0.03% solution; Device: CO2 fractional laser
- CO2 (Active Comparator): Each patient received only three CO2 fractional laser sessions 3 weeks apart
  Interventions: Device: CO2 fractional laser

INTERVENTIONS:
Drug: Bimatoprost 0.03% solution — Topical Bimatoprost 0.03% solution
  Other Names: Topical treatment of skin lesions
  Arms: Bimatoprost + CO2
Device: CO2 fractional laser — CO2 fractional laser treatment
  Other Names: laser treratment

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of combined CO2 fractional laser with Bimatoprost 0.03% as novel treatment of alopecia areata.

The main question to study is will the bimatoprost facilitate hair growth if added to fractional CO2 laser treatment in Alopecia areata.

DETAILED DESCRIPTION:
The study included 30 patients who were diagnosed clinically and dermoscopically as alopecia areata with age ranged between 16-55 years. The patients are divided into 2 groups: Group I, received fractional laser sessions with immediate and daily Bimatoprost application and Group II, received only frequent Laser sessions. Laser sessions were given to each patch once every 3 weeks, the procedure was repeated for 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Patients with alopecia areata of the scalp (multilocuolaris or single patch).
* Patient aged from 16- 55 years old in both sex.
* Other treatment wash out period is two months.

Exclusion Criteria:

* Ophiasis pattern and other patterns of alopecia areata.
* Chronic diseases of liver, heart, kidney and blood
* Pregnant women
* Infections of skin in site of intervention

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Hair regrowth | 9 weeks
  Efficacy of treatment assessed using a prognostic scoring system proposed by Mcdonald Hull and Norris for density, pigmentation, and texture of growing hair.
  Grade 1 - Regrowth of vellus hair Grade 2 - Regrowth of sparse pigmented terminal hair Grade 3 - Regrowth of terminal hair with patches of alopecia Grade 4 - Regrowth of terminal hair on scalp

SECONDARY OUTCOMES:
Side effects | 9 weeks
  The patients were asked about any side effects noticed every session by questionnaire.
  The patient satisfaction scale: - the patients were asked at final visit to rate the overall satisfaction according to whether the patient was not satisfied, slightly satisfied, satisfied or very satisfied.
  The patients were asked to report any complications as; erythema, pain, ulceration, burning sensation, ecchymosis, infection, post-inflammatory hyperpigmentation or any allergic manifestations.
Follow up assessment | 9 weeks
  The patients were followed up 3 weeks after the end of treatment sessions to detect any recurrence, complications or worsening of the lesions & final results of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- AL-Azhar University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Dhalimi MA, Al-Janabi MH, Abd Al Hussein RA. The Use of a 1,540 nm Fractional Erbium-Glass Laser in Treatment of Alopecia Areata. Lasers Surg Med. 2019 Dec;51(10):859-865. doi: 10.1002/lsm.23133. Epub 2019 Jul 18. PMID 31321800
- [Result] Choi YM, Diehl J, Levins PC. Promising alternative clinical uses of prostaglandin F2alpha analogs: beyond the eyelashes. J Am Acad Dermatol. 2015 Apr;72(4):712-6. doi: 10.1016/j.jaad.2014.10.012. Epub 2015 Jan 16. PMID 25601618
- [Result] Faghihi G, Andalib F, Asilian A. The efficacy of latanoprost in the treatment of alopecia areata of eyelashes and eyebrows. Eur J Dermatol. 2009 Nov-Dec;19(6):586-7. doi: 10.1684/ejd.2009.0766. Epub 2009 Jul 21. PMID 19620039
- [Result] El-Husseiny R, Elframawy S, Abdallah M. Comparative study between fractional carbon dioxide laser vs intralesional steroid injection in treatment of alopecia areata. Dermatol Ther. 2020 Jul;33(4):e13742. doi: 10.1111/dth.13742. Epub 2020 Jul 9. PMID 32478930
- [Result] Kim WS, Lee HI, Lee JW, Lim YY, Lee SJ, Kim BJ, Kim MN, Song KY, Park WS. Fractional photothermolysis laser treatment of male pattern hair loss. Dermatol Surg. 2011 Jan;37(1):41-51. doi: 10.1111/j.1524-4725.2010.01833.x. Epub 2010 Dec 28. PMID 21199096
- [Result] Smith S, Fagien S, Whitcup SM, Ledon F, Somogyi C, Weng E, Beddingfield FC 3rd. Eyelash growth in subjects treated with bimatoprost: a multicenter, randomized, double-masked, vehicle-controlled, parallel-group study. J Am Acad Dermatol. 2012 May;66(5):801-6. doi: 10.1016/j.jaad.2011.06.005. Epub 2011 Sep 6. PMID 21899919
- [Result] Alkhalifah A, Alsantali A, Wang E, McElwee KJ, Shapiro J. Alopecia areata update: part II. Treatment. J Am Acad Dermatol. 2010 Feb;62(2):191-202, quiz 203-4. doi: 10.1016/j.jaad.2009.10.031. PMID 20115946
- [Result] Vila TO, Camacho Martinez FM. Bimatoprost in the treatment of eyelash universalis alopecia areata. Int J Trichology. 2010 Jul;2(2):86-8. doi: 10.4103/0974-7753.77511. PMID 21712909
- [Result] Wang W, Gegentana, Tonglaga, Bagenna, Li Y. Treatment of alopecia areata with nonablative fractional laser combined with topical minoxidil. J Cosmet Dermatol. 2019 Aug;18(4):1009-1013. doi: 10.1111/jocd.12883. Epub 2019 Jun 6. PMID 31245963
- [Result] Zaher H, Gawdat HI, Hegazy RA, Hassan M. Bimatoprost versus Mometasone Furoate in the Treatment of Scalp Alopecia Areata: A Pilot Study. Dermatology. 2015;230(4):308-13. doi: 10.1159/000371416. Epub 2015 Mar 4. PMID 25765294